CLINICAL TRIAL: NCT01842542
Title: An Open-Label Study to Evaluate the Efficacy and Safety of the Neuronetics NeuroStar TMS Therapy System in Patients With Major Depressive Disorder (MDD) With Postpartum Onset.
Brief Title: Efficacy and Safety Study of NeuroStar TMS Therapy in Patients With Major Depressive Disorder With Postpartum Onset
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Neuronetics (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 44-03014-000
Record Dates: First submitted 2013-04-19; First posted 2013-04-29 (Estimated); Results first posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Depression, Postpartum
Keywords: Postpartum Depression, NeuroStar TMS Therapy, TMS
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Transcranial Magnetic Stimulation (TMS) (Experimental): Patients will receive NeuroStar Transcranial Magnetic Stimulation (TMS) therapy treatments 5 times a week for up to 8 weeks during the acute phase, 3 times during the first week, 2 times during the second week and 1 time during the third week of the taper phase.
  Efficacy Assessments will be conducted throughout the acute and taper phase at protocol specific timepoints.
  Interventions: Device: NeuroStar Transcranial Magnetic Stimulation (TMS)

INTERVENTIONS:
Device: NeuroStar Transcranial Magnetic Stimulation (TMS) — Acute phase: 120% of observed MT, 10 pulses per second, 4 second on-time, 26 second off-time, 75 trains, 3,000 total pulses/session, five times weekly for up to 8 weeks.
  3 week taper phase: 120% of observed MT, 10 pulses per second, 4 second on-time, 26 second off-time, 75 trains, 3,000 total pulses/session, 3 times during the first week, 2 times during the second week and one time during the third week. In addition to treatments, patients may receive treatment as usual at the direction of their treating physician.
  Other Names: NeuroStar TMS Therapy Treatment

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of acute NeuroStar TMS therapy in women who have postpartum depression.

DETAILED DESCRIPTION:
Evaluate the antidepressant effectiveness of acute treatment with NeuroStar TMS Therapy in patients with MDD with postpartum onset.

Determine the safety of NeuroStar TMS Therapy by assessment of any medically significant, device-related adverse events during acute treatment.

Determine the Safety of NeuroStar TMS Therapy by assessment of maternal and infant interactions on standardized bonding questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Female outpatients, 18 to 50 years of age.
* Diagnosis of DSM-IV defined Major Depressive Disorder, single or recurrent episode, with current episode duration of at least 2 weeks.
* Onset and duration of current illness within 6 months of live childbirth.
* HAMD17 total score of greater than or equal to 18 and a score on the Edinburgh Postnatal Depression scale (EPDS) greater than or equal to 10.
* Patient cannot be on an antidepressant or other psychotropic medications during the study.
* Capable and willing to provide informed consent.
* Signed HIPAA authorization.
* Able to adhere to the treatment schedule.

Exclusion Criteria:

* Individuals diagnosed by the Investigator with the following conditions (current unless otherwise stated): Depression secondary to a general medical condition, or substance-induced Seasonal pattern of depression as defined by DSM-IV;History of substance abuse or dependence within the past year(except nicotine and caffeine);Any psychotic disorder (lifetime), including schizoaffective disorder, or major depression with psychotic features in this or previous episodes;Bipolar disorder;Eating disorder (current or within the past year);Obsessive compulsive disorder (lifetime); or Post-traumatic stress disorder (current or within the past year).
* Individuals with a clinically defined neurological disorder or insult including, but not limited to:Any condition likely to be associated with increased intracranial pressure;Space occupying brain lesion;History of cerebrovascular accident;Transient ischemic attack within two years; Cerebral aneurysm; Dementia;Parkinson's disease;Huntington's chorea;Multiple sclerosis.
* History of treatment with Vagus Nerve Stimulation.
* History of failure to respond to an adequate course of ECT treatment.
* Cardiac pacemakers, implanted medication pumps, intracardiac lines, or acute, unstable cardiac disease.
* Intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed.
* Women of child-bearing potential not using a medically accepted form of contraception when engaging in sexual intercourse.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Brock, MD, Study Director — Neuronetics, Inc.
Locations (8):
- United States (8):
  - Hartford Hospital Institute of Living, Hartford, Connecticut
  - UF Health Adult Psychiatry - Springhill, Gainesville, Florida
  - Harmonex Neuroscience and Research of Pensacola, Pensacola, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Integrative Psychiatry, Louisville, Kentucky
  - TMS Medical Associates of NY, New York, New York
  - TMS Center of Lehigh Valley, Allentown, Pennsylvania
  - University of Utah - Neuropsychiatric Institute, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: TMS Treatment Sessions
Groups:
- Open Label Transcranial Magnetic Stimulation (TMS): Patients will receive NeuroStar Transcranial Magnetic Stimulation (TMS) therapy treatments 5 times a week for up to 8 weeks during the acute phase, 3 times during the first week, 2 times during the second week and 1 time during the third week of the taper phase.
  Efficacy Assessments will be conducted throughout the acute and taper phase at protocol specific timepoints.
  NeuroStar Transcranial Magnetic Stimulation (TMS): Acute phase: 120% of observed MT, 10 pulses per second, 4 second on-time, 26 second off-time, 75 trains, 3,000 total pulses/session, five times weekly for up to 8 weeks.
  3 week taper phase: 120% of observed MT, 10 pulses per second, 4 second on-time, 26 second off-time, 75 trains, 3,000 total pulses/session, 3 times during the first week, 2 times during the second week and one time during the third week. In addition to treatments, patients may receive treatment as usual at the direction of their treating physician.
Period: Overall Study
Arm/Group | Open Label Transcranial Magnetic Stimulation (TMS)
Started | 25; 36 TMS Treatment Sessions
Completed | 19; 36 TMS Treatment Sessions
Not Completed | 6; 0 TMS Treatment Sessions
Not completed — Withdrawal by Subject | 2
Not completed — Lack of Efficacy | 1
Not completed — Protocol Non-compliance | 2
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Transcranial Magnetic Stimulation (TMS): Patients will receive NeuroStar Transcranial Magnetic Stimulation (TMS) therapy treatments 5 times a week for up to 8 weeks during the acute phase, 3 times during the first week, 2 times during the second week and 1 time during the third week of the taper phase.
  Efficacy Assessments will be conducted throughout the acute and taper phase at protocol specific timepoints.
  NeuroStar Transcranial Magnetic Stimulation (TMS): Acute phase: 120% of observed MT, 10 pulses per second, 4 second on-time, 26 second off-time, 75 trains, 3,000 total pulses/session, five times weekly for up to 8 weeks.
  3 week taper phase: 120% of observed MT, 10 pulses per second, 4 second on-time, 26 second off-time, 75 trains, 3,000 total pulses/session, 3 times during the first week, 2 times during the second week and one time during the third week. In addition to treatments, patients may receive treatment as usual at the direction of their treating physician.
Arm/Group | Transcranial Magnetic Stimulation (TMS)
Number analyzed (Participants) | 25
Age, Customized [Mean (Full Range); unit: years] | 29.9 [19 to 39]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 25
EPDS Mean Baseline Score (Edinburgh Postnatal Depression Scale) [Mean (Standard Deviation); unit: units on a scale] — The EPDS is a ten-item questionnaire used for screening for postpartum depression. Total scores range from 0 to 30. Mothers who score above 10 are likely to suffer a depressive illness, while scores above 13 are likely to represent major depression. Higher score is worse outcome.
  units on a scale | 20.6 (4.15)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in EPDS Score From Baseline to End of Acute (EOA) Treatment
Description: The EPDS is a ten-item questionnaire used for screening for postpartum depression. Total scores range from 0 to 30. Mothers who score above 10 are likely to suffer a depressive illness, while scores above 13 are likely to represent major depression. Higher score at EOA means worse outcome. Once patient reached remission (EPDS<9), this was EOA treatment and scores were collected.
Time Frame: Pre to post treatment (Duration range 4 to 8 weeks)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Open Label Transcranial Magnetic Stimulation (TMS)
Number analyzed (Participants) | 19
score on a scale | -12.4 (1.769)

2. Secondary Outcome: Percentage of Patients Who Reached Remission After TMS Treatment
Description: An EPDS score less that 10 was used to indicate "remission". The 10-question Edinburgh Postnatal Depression Scale (EPDS) is a valuable and efficient way of identifying patients at risk for ³perinatal´ depression. The EPDS is easy to administer and has proven to be an effective screening tool. Mothers who score above 13 are likely to be suffering from a depressive illness of varying severity. Women are asked to answer each question in terms of the past seven days.
Time Frame: upto 8 weeks plus 3 week taper.
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Transcranial Magnetic Stimulation (TMS)
Number analyzed (Participants) | 19
Participants | 14

ADVERSE EVENTS:
Time Frame: 11 weeks
Arm/Group | Open Label Transcranial Magnetic Stimulation (TMS)
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

LIMITATIONS AND CAVEATS:
Early study termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No